CLINICAL TRIAL: NCT02990767
Title: Prediction of Early Pre-eclampsia From Maternal Factors, Biophysical and Biochemical Markers at First Trimester
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiFMIH-FMU3
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational women: collecting maternal factors, biophysical and biochemical markers at 11-13 weeks of gestation.

SUMMARY:
The aims of this study are to develop algorithms based on a combination of maternal factors, uterine artery PI, MAP and serum biomarkers to estimate patient-specific risks for early Preeclampsia (PE) and to evaluate the screening performance of such algorithms in twins.

DETAILED DESCRIPTION:
Preeclampsia (PE) is still a leading cause of fetal and maternal morbidity and mortality with an incidence of 3-5% worldwide. Despite intensive research efforts the pathogenesis of the disease is still unknown but it is likely to be multifactorial.Clinical risk factors traditionally have been used to identify women at high risk of developing preeclampsia,and biophysical factors that may help predict hypertensive disorders of pregnancy.In addition,changes in the serum concentrations of angiogenic and antiangiogenic factors are implied in the pathogenesis of PE and have possible relevance in the diagnosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* twins pregnancies delivering a phenotypically normal stillbirth or live birth at or after 24 weeks of gestation.
* twins pregnancies at at 11-14 weeks of gestation

Exclusion Criteria:

* pregnancies with major fetal abnormalities and those ending in termination, miscarriage or fetal death before 24 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twin pregnancies were recruited prospectively from women attending their routine first hospital visit in Shanghai First Maternity and Infant Hospital between December 2016 and December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Early preeclampsia | 1 year

SECONDARY OUTCOMES:
Selective intrauterine fetal growth restriction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided